CLINICAL TRIAL: NCT03891810
Title: Calm College: A Brief Mobile App Meditation Intervention Among Stressed College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Jennifer Huberty, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006896
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Stress
MeSH Terms: interventions — Calmodulin

STUDY DESIGN:
Intervention Model Description: The study design was a randomized control trial with baseline, post-intervention (8 wks from baseline), and follow-up (12 wks from baseline) assessments. College students were randomized to either a Calm College Intervention group or a delayed response group. Participants were randomized after the completion of baseline and informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calm (Experimental): The intervention ran for 8-wks with a 4-wk follow-up period. Intervention participants completed "7 days of Calm" during Week 1. For the remaining weeks (Week 2- Week 8) intervention participants were asked to meditate during the weekday from a 10-minute meditation of their choice. Throughout the intervention, the Calm College group were sent reminder texts/emails via Google Voice to participate in the meditation sessions if participants are not meditating for more than 30 minutes a week (see Participant Scripts).
  Interventions: Behavioral: Calm
- Control (No Intervention): This group was a wait list control group who received the treatment following the intervention period.

INTERVENTIONS:
Behavioral: Calm — The intervention ran for 8-wks with a 4-wk follow-up period. Intervention participants completed "7 days of Calm" during Week 1. For the remaining weeks (Week 2- Week 8) intervention participants were asked to meditate during the weekday from a 10-minute meditation of their choice. Throughout the intervention, the Calm College group were sent reminder texts/emails via Google Voice to participate in the meditation sessions if participants are not meditating for more than 30 minutes a week (see Participant Scripts).
  Arms: Calm

SUMMARY:
This research investigated the effects of a mindfulness meditation mobile application (i.e., Calm College) on reducing stress in undergraduate college students with moderate, high, or extreme levels of stress as compared to a delayed intervention group.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of a mindfulness meditation mobile application (i.e., Calm College) on reducing stress in ASU undergraduate students with moderate, high, or extreme levels of stress as compared to a delayed response group.

The study design is a randomized control trial with baseline, post-intervention (8 wks from baseline), and follow-up (12 wks from baseline) assessments. College students will be randomized to either a Calm College Intervention group or a delayed response group. Participants will be randomized after the completion of baseline and informed consent.

Aim 1: Investigate the effects of an 8-wk mobile meditation application (i.e., Calm) to reduce self-reported stress in ASU undergraduate students with moderate, high or extreme levels of stress as compared to a wait-list control group.

Aim 2: Explore the relationship between stress and reported health risk behaviors (i.e., inadequate sleep, physical inactivity, dietary behaviors, and alcohol consumption) in college students who use a mobile meditation application (i.e, Calm).

Recruitment: Participants will be recruited during September 2017. Interested participants will be directed to a Qualtrics link to complete an online eligibility screener. The screener will take approximately 10 minutes to complete (See Eligibility Survey). The survey will be free, voluntary, and available online. Participants will be allowed to skip questions in the survey.

Eligibility: Once eligibility is determined, participants will be sent an informed consent and baseline questionnaire via a Qualtrics link. This measure should take approximately 20 minutes to complete (See Informed Consent and Baseline Questionnaire). Once Informed Consent is signed and the Baseline Questionnaire is complete, participants will be randomized via an online randomizer (i.e., randomizer.com) to either a delayed response group or Calm College group. Ineligible participants will be sent an email notifying their status and given information on how to download Calm College (See Participant Scripts).

Enrollment: The Research Team will email the intervention participants that will include instructions to download Calm College (Participant Scripts). The control participants will be emailed and asked to not participate in any mindfulness based activities for 12-wks (See Participant Scrips). The intervention will run for 8-wks with a 4-wk follow-up period. Intervention participants will complete "7 days of Calm" during Week 1. For the remaining weeks (Week 2- Week 8) intervention participants will then be asked to meditate during the weekday from a 10-minute meditation of their choice. Throughout the intervention, the Calm College group will be sent reminder texts/emails via Google Voice to participate in the meditation sessions if participants are not meditating for more than 30 minutes a week (see Participant Scripts).

Tracking: Participation in the Calm College meditations will be tracked (meditation name, time of day, and time spent in meditation) by the Calm team.

Post-intervention: Post-intervention questionnaire will be emailed to intervention and control participants via a link from Qualtrics (See Post-intervention questionnaire delayed response, post-intervention questionnaire intervention). Intervention participants will have access to Calm College, but will not be asked to meditate.

Follow-up: Follow-up questionnaire will be emailed to intervention and control participants via a link from Qualtrics (See Follow-up questionnaire). Once follow-up measures have been completed, the control group will be emailed instructions on how to download Calm College.

ELIGIBILITY:
Inclusion Criteria:

* Current full-time undergraduate student at Arizona State University
* 18 years of age
* Able to read/understand English
* Own a smartphone
* A score of 14 or higher on the Perceived Stress Scale (PSS)
* Willingness to be randomized
* Willingness to download the Calm application

Exclusion Criteria:

* Participated in any mindfulness based practice within the last 6 months
* Currently utilize Calm or any other mindfulness based mobile application
* low levels of stress (i.e., less than a score of 14 assessed with the Perceived Stress Scale)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Stress (Perceived Stress Scale (PSS) score) | 8 weeks post baseline
  The PSS is a 10-item inventory used for the assessment of perceived stress. The scale measures the degree to which situations are appraised as stressful. ?". The items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Higher scores indicate higher levels of stress. Scores are computed via sum.

SECONDARY OUTCOMES:
Sleep (Self-reported sleep using the Patient-Reported Outcomes Measurement Information System Short Form (PROMIS 8a)) | 8 weeks post baseline
  The PROMIS short-from is an 8-item inventory used to assess sleep disturbance in adults. The first seven questions follow the same pattern and are rated on a 5-point Likert scale ranging from 1 (Not at all) to 5 (Very much). The last question is rated on a reversed 5-point Likert scale ranging from 5 (Very poor) to 1 (Very good).
Physical Activity (Aerobic and strength training, using the Youth Risk Behavior Survey (YRBS)) | 8 weeks post baseline
  The YRBS is 99-item survey that assesses six categories of priority health-risk behaviors among youth and young adults, however only the sub-scale for physical activity was assessed for this outcome. Higher scores indicate higher levels of physical activity. There are 10 items in this sub scale, and scores range from 0-10. Scored are computed via sum of questions.
Diet (Fruit and vegetable consumption, using the Youth Risk Behavior Survey (YRBS)) | 8 weeks post baseline
  The YRBS is 99-item survey that assesses six categories of priority health-risk behaviors among youth and young adults, however only the sub-scale for diet was assessed for this outcome. Higher scores indicate higher levels of fruit and vegetable consumption. There are 20 items on this sub scale, and scores range from 0-20. Scored are computed via sum of questions.
Alcohol Consumption (Alcohol consumption, using the Youth Risk Behavior Survey (YRBS)) | 8 weeks post baseline
  The YRBS is 99-item survey that assesses six categories of priority health-risk behaviors among youth and young adults, however only the sub-scale for alcohol consumption was assessed for this outcome. Higher scores indicate higher levels of alcohol consumption. There are 6 items on this sub scale and scored range from 0-6. Scored are computed via sum of questions.
Five Factor Mindfulness Questionnaire (FFMQ) | 8 weeks post baseline
  The FFMQ is a 39-item self-report inventory used for the assessment of multiple constructs of mindfulness skills. The inventory assesses five subscales: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. The response items are rated on a 5-point Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true). The facet scores range from 8-40 with the exception of non-reactivity to inner experience which ranges from 7-35. Higher scores indicate higher levels of mindfulness.
Self-Compassion Survey Short-Form (SCS-SF) | 8 weeks post baseline
  The SCS-SF is a 12-item survey assessing three subscales: self-kindness versus self-judgment, common humanity versus isolation, and mindfulness versus over-identification. The response items are rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Higher scores indicate higher levels of self-compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baum A. Stress, intrusive imagery, and chronic distress. Health Psychol. 1990;9(6):653-75. doi: 10.1037//0278-6133.9.6.653. PMID 2286178
- [Background] Edenfield TM, Saeed SA. An update on mindfulness meditation as a self-help treatment for anxiety and depression. Psychol Res Behav Manag. 2012;5:131-41. doi: 10.2147/PRBM.S34937. Epub 2012 Nov 23. PMID 23175619
- [Background] Leppink EW, Odlaug BL, Lust K, Christenson G, Grant JE. The Young and the Stressed: Stress, Impulse Control, and Health in College Students. J Nerv Ment Dis. 2016 Dec;204(12):931-938. doi: 10.1097/NMD.0000000000000586. PMID 27575792
- [Background] McIndoo CC, File AA, Preddy T, Clark CG, Hopko DR. Mindfulness-based therapy and behavioral activation: A randomized controlled trial with depressed college students. Behav Res Ther. 2016 Feb;77:118-28. doi: 10.1016/j.brat.2015.12.012. Epub 2015 Dec 23. PMID 26745622
- [Background] Caldwell K, Harrison M, Adams M, Quin RH, Greeson J. Developing mindfulness in college students through movement-based courses: effects on self-regulatory self-efficacy, mood, stress, and sleep quality. J Am Coll Health. 2010 Mar-Apr;58(5):433-42. doi: 10.1080/07448480903540481. PMID 20304755
- [Derived] Huberty J, Green J, Glissmann C, Larkey L, Puzia M, Lee C. Efficacy of the Mindfulness Meditation Mobile App "Calm" to Reduce Stress Among College Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 25;7(6):e14273. doi: 10.2196/14273. PMID 31237569